CLINICAL TRIAL: NCT00687089
Title: Examination of Cognitive Function, Weight, Sexual Function in Patients Receiving Treatment With Subutex at 3 Months Without Using Opiates
Brief Title: Examination of Cognitive Function in Patients Treated With Subutex
Status: Completed | Type: Observational
Sponsor: BeerYaakov Mental Health Center (Other Government)
Collaborators: Ebetim Clinic (Other)
Responsible Party: Aviva Wolf, "Hebetim" psychiatric and psychologic clinic- private clinic
Other Study IDs: Subutex-214CTIL
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Opiate Addiction
Keywords: Opiates; Subutex; Buprenorphine; Patients who addicted to opiates
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subutex group: People who used opiates and willing to start with subutex treatment
  Interventions: Other: Sexual, cognitive functional tests and measurement weight

INTERVENTIONS:
Other: Sexual, cognitive functional tests and measurement weight

SUMMARY:
People who addicted to Heroin and other opiates suffer from a disease with approved genetic basis. It causes to a behavioral response as searching and using those drugs even though they know it causes severe damages as physiological, familiar and legal affairs.

The popular treatment's goal is to "clean" the people from any drug. In a medical and pharmacological point of view there is no sense in this approach for all people. This point of view believes that Buprenorphine (Subutex) is a correct pharmacological treatment.

The hypothesis of this research is that people using Buprenorphine have difficulties in gaining weight, in sexual and cognitive function (according to subjects' reports)

DETAILED DESCRIPTION:
People who addicted to Heroin and other opiates suffer from a disease with approved genetic basis. It causes to a behavioral response as searching and using those drugs even though they know it causes severe damages as physiological, familiar and legal affairs.

The popular treatment's goal is to "clean" the people from any drug. In a medical and pharmacological point of view there is no sense in this approach for all people. This point of view believes that Buprenorphine (Subutex) is a correct pharmacological treatment.

The hypothesis of this research is that people using Buprenorphine have difficulties in gaining weight, in sexual and cognitive function (according to subjects' reports) We examine people who stopped opiates and began Buprenorphine. Every participant in the study will have two visits: the first one before receiving Buprenorphine and the second one after 3 months of receiving Buprenorphine.

ELIGIBILITY:
Inclusion Criteria:

* People who suffer from addiction problems (opiates)
* People who willing to to start Buprenorphine treatment
* People who willing to cooperate with study tests and questionnaires
* People aged 18 to 70

Exclusion Criteria:

* People who suffer from any neurocognitive problems
* People who suffer from mental illnesses
* People who are having legal guardian

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who suffer from addiction problems (opiates) and willing to start Buprenorphine treatment
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
ASI quationarry, neurocognitive computerized tests, MMSE test, Sexual function questionnaire and satisfaction questionnaire | In 2 visits during the study

REFERENCES:
- See also: "Ebetim" clinic where the study will be conducted — http://www.ebetim.co.il